CLINICAL TRIAL: NCT05017298
Title: Clinical Study for Subjects With Coronavirus 2019 (COVID-19) Using Multiple Dose Intravenous Infusions of Allogeneic Adipose Tissue-Derived Mesenchymal Stem Cells (AdMSCs)
Brief Title: Clinical Study for Subjects With COVID-19 Using Allogeneic Adipose Tissue-Derived Mesenchymal Stem Cells
Acronym: AdMSCs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Celltex Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTX0020-004
Record Dates: First submitted 2021-08-18; First posted 2021-08-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-04

CONDITIONS: Corona Virus Infection; Covid19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: The Phase 2 study is a randomized, double blind and placebo control study conducted initially in a single clinic facility.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Each subject receives three separate doses of 200 million allogeneic adipose-derived mesenchymal stem cells via intravenously infusion on days 0, 3, and 6 with a total of 600 million AdMSCs during 7 days in addition to their standard of care.
  Interventions: Biological: Allogeneic adipose-derived stem cells
- Control Group (Placebo Comparator): The control group will receive placebo infusion on day 0, 3 and 6 along with standard of care.
  Interventions: Biological: Allogeneic adipose-derived stem cells

INTERVENTIONS:
Biological: Allogeneic adipose-derived stem cells — Culture expanded mesenchymal stem cells isolated from a patient's own abdominal fat tissue
  Other Names: Celltex-AdMSCs

SUMMARY:
This is an interventional new drug clinical trial for a Phase 2 randomized, double-blind, and placebo control study using intravenous injection of allogeneic adipose stem cells (Celltex AdMSCs) for subjects with severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years.
* Male and female
* Must understand and voluntarily sign an Informed Consent for study participation obtained prior to undergoing any study-specific procedures
* Diagnosed as COVID-19 based upon SARS-CoV-2 RT-PCR test positive
* Clinical diagnosis meets severe and/or critical parameters
* Male participants must be willing to ensure their partners do not become pregnant either by practicing abstinence or the use of condoms during sexual activity

Exclusion Criteria:

* Participation in another clinical study (with use of another Investigational Medical Product) within 3 months prior to study treatment start
* Unwillingness or inability to comply with study procedures
* Patients with serious basic diseases that affect survival, including blood diseases, cachexia, active bleeding, severe malnutrition, etc.
* Clinically active malignant disease
* Subjects who are receiving ECMO and CRRT currently
* History of known pulmonary embolism or known secondary anti-phospholipid syndrome
* Known or suspected hypersensitivity to any components used to culture the AdMSCs, e.g. BSA and sulfur containing products (e.g., DMSO)
* Known or suspected allergic to diphenhydramine.
* Major trauma or surgery within 14 days of study treatment start
* Mental condition rendering the subject (or the subject's legally acceptable representative[s]) unable to understand the nature, scope and possible consequences of the study
* Alcohol, drug, or medication abuse within one year prior to study treatment start
* Any condition that, in the Investigator's opinion, is likely to interfere with evaluation of the AdMSC therapy or satisfactory conduct of the study
* Irreversible severe end organ failure, such as heart failure/attack, stroke, liver and renal failure due to other disease conditions
* Patients or family history with hypercoagulable status, such as protein C/protein S deficiency, factor V Leiden, prothrombin gene mutation, dysfibrinogenemia, etc.
* History of long-term use of immunosuppressive agents
* Organ transplants in the past 6 months
* Pregnant, breastfeeding, or desire to become pregnant or unwilling to practice birth control during participation in the study duration, unless surgically sterilized or postmenopausal during the study.
* Patients with previous pulmonary obstructive pneumonia, severe pulmonary interstitial fibrosis, alveolar proteinosis, allergic alveolitis, and other known viral pneumonia or bacterial pneumonia before COVID-19 infection. The pulmonary imaging revealed the interstitial damage of lungs before the COVID-19 confirmed.
* QT interval shows greater than 450 ms in males and 470 ms in females in the medical histories or during screen EKG test.
* Subjects are not medically unstable at time of infusion including but not limiting unstable hypertension, pulse, oximetry, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Safety of AdMSC injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study based on the rate of all AdMSC-associated adverse events (AEs) in all subjects. | 6 months
  Incidence of treatment-related adverse events and severe adverse events during the study period
Safety for AdMSCs based upon incidence of all AEs | 6 months
  Grouped by Medical Dictionary for Regulatory Activities (MedDRA)
Compare the mortality rate | 6 months
  AdMSC treating group vs. control group

SECONDARY OUTCOMES:
Recognized immune measurements evaluating patients' symptom changes and overall function | 6 months
  To evaluate change of sequential organ failure assessment (SOFA) score as compare to the baseline
Organ functional tests including blood specific enzymes and proteins | 6 months
  To evaluate the efficacy of allogeneic AdMSCs for COVID-19
Duration (days) of weaning from mechanical ventilation | 6 months
  Compared to control group
Duration (days) of ICU monitoring | 6 months
  Compared to control group
Duration (days) of vasoactive agent's usage | 6 months
  Compared to control group
Duration of hospitalization (days) | 6 months
  Compared to control group
Proportions of SARS-CoV-2 RT-PCR change to negative from respiratory tract specimens (oropharyngeal swabs) using CDC standard method | 6 months
  Compared to control group
Proportions of quantifying viral RNA in stool change to negative in final follow-up using CDC standard method | 6 months
  Compared to control group
Proportions of blood SARS-CoV-2 antibodies IgM/IgG show positive | 6 months
  Compared to control group

OTHER OUTCOMES:
Mortality rate down to 0% | 6 months
  For severe and critical cases
Achieve at least 30% more proportion of severe patients in AdMSC study group without developing organ failure or recovery from previous organ failure | 6 months
  Compared to control group

CONTACTS AND LOCATIONS:
Overall Officials: Derek W Guillory, MD, Principal Investigator — Root Causes Medicine